CLINICAL TRIAL: NCT01076166
Title: A Multi-center, Post-Marketing Observational Study to Identify the Recovery Time in Children With Lower Respiratory Tract Infections Treated With Klacid Granules for Oral Suspension.
Brief Title: Recovery Time in Children With Lower Respiratory Tract Infections Treated With Klacid® Granules for Oral Suspension.
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Savary Om/ Regional Medical Director, Abbott Laboratories
Other Study IDs: P10-813
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2011-03-07 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Lower Respiratory Tract Infection
Keywords: Post-marketing observational study; Lower respiratory tract infections; Klacid Granules for Oral Suspension
MeSH Terms: interventions — Clarithromycin; Suspensions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with lower respiratory tract infection: Thai children with lower respiratory tract infections on Klacid Granules for Oral Suspension
  Interventions: Drug: clarithromycin (Klacid) granules for oral suspension

INTERVENTIONS:
Drug: clarithromycin (Klacid) granules for oral suspension — clarithromycin (Klacid) Granules for Oral Suspension
  Other Names: clarithromycin; Klacid Granules for Oral Suspension; Biaxin XL

SUMMARY:
Klacid Granules for Oral Suspension provides short symptoms' recovery time in Thai children with lower respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower respiratory tract infection.
* Patient is male or female > 6 months and < 12 years of age.
* Prescription of Klacid Granules for Oral Suspension is at the discretion of the investigators according to the clinical condition of the patients
* Patients who are suitable for treatment with Klacid Granules for Oral Suspension according to the Prescribing Information

Exclusion Criteria:

* Known hypersensitivity to or previously intolerant of macrolides.
* Illness severe enough to warrant hospitalization or parenteral therapy.
* Concomitant use of any of the following medications:

  * Drugs metabolized by CYP3A isozyme: alprazolam, astemizole, carbamazepine, cilostazol, cisapride, cyclosporin, disopyramide, ergot alkaloids, lovastatin, methylprednisolone, midazolam, omeprazole, oral anticoagulants (e.g. warfarin), pimozide, quinidine, rifabutin, sildenafil, simvastatin, tacrolimus, terfenadine, triazolam and vinblastine.
  * Drugs metabolized by other isozymes within CYP450 system: phenytoin, theophylline and valproate.
  * Colchicine
  * Digoxin
  * Ritonavir.
* Severe immunodeficiency and chronic disease conditions.
* Renal or hepatic impairment.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Out-patients in Thailand
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Savary Om, M.D., Study Director — Abbott
Locations (16):
- Thailand (16):
  - Site Reference ID/Investigator# 27424, Bangkok
  - Site Reference ID/Investigator# 46824, Bangkok
  - Site Reference ID/Investigator# 16261, Bangkok
  - Site Reference ID/Investigator# 46825, Bangkok
  - Site Reference ID/Investigator# 27428, Bangkok
  - Site Reference ID/Investigator# 27425, Bangkok
  - Site Reference ID/Investigator# 27423, Bangkok
  - Site Reference ID/Investigator# 27426, Bangkok
  - Site Reference ID/Investigator# 46823, Chiang Mai
  - Site Reference ID/Investigator# 27434, Chumphon
  - Site Reference ID/Investigator# 27433, Chumphon
  - Site Reference ID/Investigator# 27431, Nakhon Ratchasima
  - Site Reference ID/Investigator# 27441, Nong Khai
  - Site Reference ID/Investigator# 27429, Phitsanulok
  - Site Reference ID/Investigator# 27432, Rayong
  - Site Reference ID/Investigator# 27430, Samutsakorn

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 337 participants were enrolled in the study. 308 were analyzed as 29 participants had protocol deviations: Took Klacid less than 5 days (9), took Klacid more than 14 days (4), Klacid intravenous formulation used instead of granules (9), participants enrolled prior to signed study agreement (5), and age less than 6 months (2).
Groups:
- Klacid Granules (Total): Male or female Thai children more than 6 months and less than 12 years of age with lower respiratory tract infections treated with Klacid (clarithromycin) Granules for Oral Suspension according to the Prescribing Information.
Period: Overall Study
Arm/Group | Klacid Granules (Total)
Started | 337
Completed | 328
Not Completed | 9
Not completed — Adverse Event | 3
Not completed — Symptoms improved/resolved | 6

BASELINE CHARACTERISTICS:
Groups:
- Klacid Granules (Total): The per-protocol population (308 participants) of male or female Thai children more than 6 months and less than 12 years of age with lower respiratory tract infections treated with Klacid (clarithromycin) Granules for Oral Suspension according to the Prescribing Information.
Arm/Group | Klacid Granules (Total)
Number analyzed (Participants) | 308
Age Continuous [Median (Full Range); unit: years] — Based on per protocol population (308 participants).
  years | 4.2 [0.50 to 11.90]
Age, Customized [Number; unit: participants] — Based on per protocol population (308 participants).
  participants
    > 6 months to 3 years | 80
    Between 3 and 5 years | 118
    > 5 and < 12 years | 110
Sex: Female, Male [Count of Participants; unit: Participants] — Based on per protocol population (308 participants).
  Participants
    Female | 147
    Male | 161
Region of Enrollment [Number; unit: participants] — Based on per protocol population (308 participants).
  participants
    Thailand | 308
Diagnosis [Number; unit: participants] — Participant diagnosis at study entry for the per protocol population (308 participants).
  participants
    Bronchitis | 278
    Pneumonia | 30
Risk Factor--Upper Respiratory Tract Infections [Number; unit: participants] — The frequency in which participants had experienced upper respiratory tract infections (URTI) in the past, for the per protocol population (308 participants).
  participants
    URTI 1 to 2 times per year | 98
    URTI 3 to 6 times per year | 76
    URTI 7 to 10 times per year | 5
    URTI > 10 times per year | 0
    URTI not reported | 129
Risk Factor--Lower Respiratory Tract Infections [Number; unit: participants] — The frequency in which participants had experienced lower respiratory tract infections (LRTI) in the past, for the per protocol population (308 participants).
  participants
    LRTI 1 to 2 times per year | 111
    LRTI 3 to 6 times per year | 27
    LRTI 7 to 10 times per year | 9
    LRTI > 10 times per year | 0
    LRTI not reported | 161

OUTCOME MEASURES:

1. Primary Outcome: Average Time From Baseline to Recovery From Fever and Other Symptoms
Description: Participants were observed during his/her Klacid treatment (5 to 14 days). A medical appointment was made 6 to 14 days after the first visit. Participants' symptoms were rated using one of the following categories: resolved, improved, not changed, or worse. Associated dates were also recorded. Symptoms included, but were not limited to, fever, cough, chest/abdominal pain, and vomiting. Recovery was defined as the disappearance of all signs and symptoms of infection.
Time Frame: Baseline to 14 days
Population: A total of 29 patients were excluded for protocol deviations: Took Klacid less than 5 days (9), took Klacid more than 14 days (4), Klacid intravenous formulation used instead of granules (9), participants enrolled prior to signed study agreement (5), and age less than 6 months (2). Average time to recovery was based on 171 recovered patients.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Klacid Granules (Total Number Recovered): Male or female Thai children more than 6 months and less than 12 years of age with lower respiratory tract infections treated with Klacid (clarithromycin) Granules for Oral Suspension according to the Prescribing Information who were in the recovered population.
- Klacid Granules (Bronchitis, Recovered): Participants in the recovered population who had a diagnosis of bronchitis at study entry.
- Klacid Granules (Pneumonia, Recovered): Participants in the recovered population who had a diagnosis of pneumonia at study entry.
Arm/Group | Klacid Granules (Total Number Recovered) | Klacid Granules (Bronchitis, Recovered) | Klacid Granules (Pneumonia, Recovered)
Number analyzed (Participants) | 171 | 163 | 8
Days | 7.18 (2.33) | 7.14 (2.35) | 7.88 (1.81)

2. Secondary Outcome: Number and Type of Adverse Events
Description: Adverse events were collected during the course of the study up to 30 days or 5 half-lives following the last dose of Klacid. The number of participants experiencing a serious or non-serious adverse event are summarized. See the Reported Adverse Event section for details.
Time Frame: Baseline to 14 days
Population: The safety population included all participants who took at least 1 dose of Klacid.
Measure: Number; unit: Participants
Arm/Group | Klacid Granules (Total)
Number analyzed (Participants) | 337
Participants
  Serious adverse events | 2
  Non-serious adverse events | 1

ADVERSE EVENTS:
Time Frame: All adverse events that occurred during the course of the study were reported in detail on case report forms. Adverse events occurring during the study were reported up to 30 days or 5 half-lives after the last dose of Klacid.
Description: The 6 serious adverse events that occurred in 2 participants and the one non-serious adverse event are summarized.
Arm/Group | Klacid Granules (Total)
Serious Adverse Events (participants affected / at risk) | 2/337
Other Adverse Events (participants affected / at risk) | 1/337
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Klacid Granules (Total) (N=337)
Drug ineffective (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Klacid Granules (Total) (N=337)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.